CLINICAL TRIAL: NCT07082010
Title: A Novel Digital Platform for Measurement-based Peer Supervision of Non-specialist Providers Conducting Brief Psychological Interventions
Brief Title: Measurement-Based Peer Supervision App for Non-Specialist Providers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dimagi Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Harvard Medical School (HMS and HSDM) (Other); Baylor Scott and White Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R44MH130305 (NIH); 2R44MH130305-02 (NIH)
Record Dates: First submitted 2025-05-14; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Training of Mental Health Professionals; Training of Frontline Health Workers
Keywords: anxiety; depression; behavioral activation; task-sharing; community health workers; digital health
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBPS App (Experimental): Study participants (i.e., non-specialist providers) will use a web application to support measurement-based peer supervision (MBPS) activities (e.g., rating and reviewing therapy sessions) performed with standardized patients in mock scenarios
  Interventions: Device: MBPS App

INTERVENTIONS:
Device: MBPS App — A MBPS web application designed and built on a customizable case management platform (CommCare) to support non-specialist providers will be used by study participants for approximately 3 months.

SUMMARY:
The goal of this project is to enhance and evaluate the efficacy of a scalable digital solution designed to help train and support the work of non-specialist providers (NSPs), such as community health workers, to deliver therapy to individuals with anxiety and/or depression. The main questions this project aims to answer are:

* Can a digital tool help NSPs feel more confident in counseling patients?
* How can a digital tool be designed to optimally support the work of NSPs?

DETAILED DESCRIPTION:
There is a critical shortage of mental health specialists (i.e., psychiatrists, psychologists, licensed mental health counselors) and a growing mental health crisis in the US. Task sharing, whereby highly qualified health workers share specific tasks non-specialist providers (NSPs) with less training and fewer qualifications in order to make more efficient use of the available human resources, is an approach that can scale and address unmet mental health needs, particularly in hard-to-reach communities with limited to no access to specialist care. The investigators propose a comprehensive solution to support a task sharing approach for delivering high quality brief psychosocial interventions. Our proposed digital platform is designed to support measurement-based peer supervision (MBPS), which includes the ability for NSPs to record therapy sessions, rate them using a validated quality scale, and review ratings safely and securely with peers in moderated group discussions. The investigators developed and successfully demonstrated acceptability, usability, and potential feasibility of digitally-enabled MBPS to support NSP performance and quality of care in Phase I. The goal of this Phase II project is to enhance and evaluate the efficacy of this digitally-enabled MBPS tool with NSPs working directly in communities. The investigators will address this goal with three specific aims.

In Aim 1, the investigators will build an enhanced version of the digital platform based on Phase I feedback and direct input from NSPs.

In Aim 2, the investigators will conduct a mixed methods evaluation of digitally-enabled MBPS with 50 target end users, i.e., NSPs recruited from a large health system in Texas and recently trained in behavioral activation. During this period, NSPs will engage in mock sessions with standardized patients. Primary outcomes of interest will be NSP session quality in delivering behavioral activation therapy and counselor self-efficacy.

Results of this Phase II work can provide important insights to guide the implementation and scaling of effective delivery of psychosocial interventions and program quality improvement, with the long-term goal of improving mental health outcomes in hard-to-reach communities that can benefit the most from NSP-led support.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* English-speaking; and
* Completed EMPOWER Behavioral Activation training

Exclusion Criteria:

- Unable to participate in virtual meetings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioral Activation (BA) Quality over Sessions | 12 weeks, from enrollment to study completion (assessed every 4 weeks)
  The BA Quality Scale for Healthy Activity Program score will be used to assess differences in BA quality over 3 sessions as scored by self, peer, and expert based on review of recordings. The BA Quality Scale ranges from 0 to 8, with higher scores indicating higher quality.
Change in Self-Efficacy | 12 weeks, from enrollment to study completion (assessed at Baseline and Endline)
  The Counselor Self-Efficacy Scale (SE-12) will be used to assess change in self-efficacy before and after the intervention. The scale ranges from 0 to 120 with higher scores indicating higher self-efficacy.

SECONDARY OUTCOMES:
System Usability | End of 12 weeks, at study completion
  The Positive System Usability Scale (SUS) will be assessed at the end of the intervention period to assess perceived usability of the intervention. The scale ranges from 0 to 100, with higher scores indicating higher usability.
System User Satisfaction | End of 12 weeks, at study completion
  The Net Promoter Score (NPS) will be used to assess user satisfaction with the intervention. The NPS is 1 item with a score ranging from -100 to 100, with higher scores indicating higher user satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Xian Ho, PhD, Principal Investigator — Dimagi Inc.
Locations (1):
- Baylor Scott & White Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data; results will ll be reported in aggregate.

REFERENCES:
- [Background] Poudyal A, Lewis DM, Taha S, Martinez AJ, Magoun L, Ho YX, Carmio N, Naslund JA, Sanchez K, Lesh N, Patel V. Designing an App to Support Measurement-Based Peer Supervision of Frontline Health Workers Delivering Brief Psychosocial Interventions in Texas: Multimethod Study. JMIR Form Res. 2024 Mar 11;8:e55205. doi: 10.2196/55205. PMID 38466971